CLINICAL TRIAL: NCT05725720
Title: Role of the Gut Microbiome in the Outcome of Diffuse Large B-Cell Lymphoma Patients Treated With CAR-T Cell Therapy
Acronym: MicroCar
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Pier Luigi Zinzani, Full Professor of Hematology, University of Bologna
Other Study IDs: IG2022id27350
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Gut microbiome; CAR T-cell therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gut microbiome analysis — Characterization of the compositional and functional modifications of gut microbiome in patients affected by lymphoma undergoing therapy with CAR-T cells from baseline until the restaging after 18 months from the CAR-T cell infusion

SUMMARY:
Despite impressive outcomes in selected patients, significant heterogeneity in clinical response to CAR-T cell therapy remains. The gut microbiome (GM) has recently emerged as one of the key modifiable factors of prognosis and response to treatment in cancer patients, with high-diversity profiles rich in health-associated taxa while poor in pathobionts generally associated with better response and longer survival. Currently, it is unknown if GM also modulates anti-tumor responses to CAR-T cells and related toxicities in lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients affected by histologically confirmed DLBCL.
3. Patients amenable for CAR-T cell therapy as for clinical approved indication (commercial products).
4. Patients must provide written informed consent.

Exclusion Criteria:

1. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results.
2. Concurrent second malignancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 90 relapsed/refractory diffuse large B-cell lymphoma adult (≥18 years) patients undergoing CAR-T cell therapy will be enrolled over 3 years, treated and followed up with fecal sample collection until 18 months after CAR-T cell infusion.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of GM heterogeneity (taxa) in diffuse large B-cell lymphoma patients undergoing CAR-T cell therapy. | 24 months
  Characterization of the compositional and functional modifications of GM in patients affected by lymphoma undergoing therapy with CAR-T cells from baseline until the restaging after 18 months from the CAR-T cell infusion. GM profiling will be achieved by next-generation sequencing approaches, including 16S rRNA gene-based sequencing for diversity and compositional structure, and shotgun metagenomics for species-level and functional insights, including information on eukaryotes and viruses.

SECONDARY OUTCOMES:
Correlation between GM and CAR-T cell therapy outcomes in terms of response, toxicity and disease control. | 4 years
  Define novel GM signatures that relate to more favorable response to the CAR-T treatment and/or reducing the occurrence of side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Of Hematology "Seràgnoli", Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided